CLINICAL TRIAL: NCT03383107
Title: Effect of Radiotherapy Variables on Circulating Effectors of Immune Response and Local Microbiome
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: 1708018471
Record Dates: First submitted 2017-12-13; First posted 2017-12-26 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimens will be collected prospectively from consented patients at baseline, during radiation therapy, at completion of radiation therapy and during 3-4 month follow up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1a - Prostate Cancer: Standard fractionation RT to 81 Gy in 45 fx over 9 weeks
- Cohort 1b - Prostate Cancer: Hypofractionated RT to 36.25 Gy in 5 fx over 1-2 weeks
- Cohort 2a - Breast cancer: Standard fractionation breast and nodal RT to 50 Gy in 25 fx over 5 weeks
- Cohort 2b - Breast Cancer (Partial Breast ): Partial breast RT to 30 Gy in 5 fx over 2 weeks

SUMMARY:
Exposure to radiation can impact immune cells that are present in the blood, such as lymphocytes. It is hypothesized that larger radiation fields and/or longer courses of radiation, result in greater decrease in immune cells. To test this hypothesis, investigators will take blood samples from subjects undergoing two different standard of care radiation regimens for prostate cancer, and subjects undergoing two different standard of care regimens for breast cancer.

DETAILED DESCRIPTION:
The study prospectively collects blood specimens for assessment of peripheral immune mediators in 4 distinct clinical settings of standard radiotherapy. In addition to collecting blood specimens, the study will also collect physical and dosimetric information of treatment such as total dose, number of treatments, and/or size of the radiation targe, as these will allow the investigators to study the impact of radiation variables on the immune system. Stool specimens will be collected at baseline, end of radiation therapy and during the follow up visit to detect microbiome changes associated with different radiation treatment at various time points. Humans are colonized by commensal bacteria, which outnumber human cells. These normal bacteria colonize mucosal surfaces and play a critical role in immunity. It is hypothesized that the underlying microbiota may also undergo changes in composition that correspond to the regimen of radiation that is utilized. By collecting stool specimens, investigators will be able to study microbial changes and how these changes correlate with alteration in immune mediators (i.e., lymphocytes, cytokines) present in blood samples before, during and after radiation; and explore the association between these parameters and type of radiation received.

ELIGIBILITY:
Cohort 1a and b: Prostate cancer subjects undergoing 9 week radiation

Inclusion criteria:

* Biopsy-proven diagnosis of prostate adenocarcinoma
* Age ≥ 18

Exclusion criteria:

* History of prior pelvic radiation (external beam or brachytherapy)
* Prior or concurrent lymphomatous/hematogenous malignancy, or history of prior/concurrent invasive malignancy during the past 5 years
* History of hormone therapy such as LHRH agonists (gosrelin, leuprolide), anti-androgens (flutamide, bicalutamide), surgical castration (orchiectomy)
* History of irritable bowel disease
* Evidence of lymph node involvement or metastatic disease

Cohort 2a : Breast cancer subjects undergoing standard fractionation RT of 5 weeks

Inclusion criteria:

* Biopsy-proven diagnosis of invasive breast cancer, s/p breast surgery to negative margins, and requiring adjuvant breast and nodal RT
* Age ≥ 18

Exclusion criteria:

* History of prior radiation therapy to the ipsilateral breast
* Prior or concurrent lymphomatous/hematogenous malignancy, or history of prior/concurrent invasive malignancy during the past 5 years
* < 1 month from completion of chemotherapy to start of RT
* Evidence of metastatic disease

Cohort 2b: Breast cancer subjects undergoing PBI

Inclusion criteria:

* Post-menopausal women defined as either 1) at least 2 years without menstrual period or 2) or patients older than 50 with serological evidence of post-menopausal status or 3) hysterectomized patients of any age with FSH confirmation of post-menopausal status.
* Post-segmental mastectomy with negative margins
* If bilateral, pT1 breast cancer, excised with negative margins AND/OR
* pTis excised with negative margins
* Clinically N0 or pN0 or sentinel node negative
* Diagnosis of ductal carcinoma in situ DCIS, limited to <2cm size of DCIS and to lesions of low or intermediate grade, excised (or re-excised) with final negative margins ( no DCIS on inked margins).
* Age ≥ 18

Exclusion criteria:

* History of prior radiation therapy to the ipsilateral breast
* Presence of a proportion of DCIS in the core biopsy specimen which is compatible with extensive intraductal component (EIC).
* < 1 month from completion of chemotherapy to start of RT
* Evidence of metastatic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with biopsy-proven, non-metastatic prostate adenocarcinoma, meeting the inclusion/exclusion criteria below, and electing to undergo definitive radiation treatment, will be eligible for participation.
  Women with biopsy-proven, non-metastatic invasive or in situ breast cancer meeting the inclusion/exclusion criteria below will be eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
prospectively collecting blood specimens to assess peripheral immune mediatiors in 4 distinct clinical settings | 4 years
  prospectively collect collect physical and dosimetric information of treatment and sequential blood samples for assessment of peripheral immune mediators in 4 distinct clinical settings of standard radiotherapy (2 for breast and 2 for prostate cancer)
distribution and frequency of peripheral immune mediators before, during and after radiotherapy will be assessed from blood samples that are collected at various time points | 4 years
  To characterize the distribution and frequency of peripheral immune mediators before, during and after radiotherapy in each of the 4 subsets of the prospective trial.

SECONDARY OUTCOMES:
microbiome changes associated with different radiation treatments through collection of stool microbiome samples at different time points | 4 years
  explore microbiome changes associated with different radiation treatments through collection of stool microbiome samples at baseline, at the end of radiation therapy, and during follow up after completion of Radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Formenti SC, Demaria S. Combining radiotherapy and cancer immunotherapy: a paradigm shift. J Natl Cancer Inst. 2013 Feb 20;105(4):256-65. doi: 10.1093/jnci/djs629. Epub 2013 Jan 4. PMID 23291374
- [Background] Formenti SC, Demaria S. Radiation therapy to convert the tumor into an in situ vaccine. Int J Radiat Oncol Biol Phys. 2012 Nov 15;84(4):879-80. doi: 10.1016/j.ijrobp.2012.06.020. No abstract available. PMID 23078897